CLINICAL TRIAL: NCT04863222
Title: Clinical and Radiographic Success of Mineral Trioxide Aggregate (MTA) vs Septodont Biodentine in Primary Molars in Pulpotomy and Indirect Pulp Cap Treatments
Brief Title: Clinical and Radiographic Success of MTA vs Biodentine
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0994
Record Dates: First submitted 2021-03-15; First posted 2021-04-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Indirect Pulp Cap; Pulpotomy
MeSH Terms: interventions — mineral trioxide aggregate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MTA, then Biodentine (Experimental): The participant will receive the standard of care procedure using MTA in on a right primary molar. A left primary molar will then be treated using Biodentine.
  Interventions: Device: Biodentine; Biological: mineral trioxide aggregate (MTA)
- Biodentine, then MTA (Experimental): Investigators will prepare and treat a participants right primary molar with Biodentine. The participant will then receive the standard of care procedure using MTA in on a left primary molar.
  Interventions: Device: Biodentine; Biological: mineral trioxide aggregate (MTA)

INTERVENTIONS:
Device: Biodentine — During a patients procedure, one tooth will receive Biodentine instead of MTA.
Biological: mineral trioxide aggregate (MTA) — mineral trioxide aggregate (MTA)

SUMMARY:
The purpose of this prospective study is to compare the clinical and radiographic success of MTA and Biodentine as a medicament in vital pulp therapy in maxillary and mandibular primary molars in a pediatric population. There is limited research currently on Biodentine since it's a novel product. Biodentine is less expensive than MTA and does not cause discoloration like MTA. Biodentine may be an alternative medicament used for vital pulp therapy in primary molars.

DETAILED DESCRIPTION:
This is a interventional randomized split mouth prospective study that evaluates the clinical and radiographic success of mineral trioxide aggregate (MTA) and Biodentine as pulpotomy and indirect pulp cap (IPC) medicaments. Male and female participants ages two to twelve who need at least two quadrants of treatment will be enrolled in the trial. Participants will be treated at Geisinger Medical Center, Danville, and Geisinger Bloomsburg Hospital operating rooms for full mouth rehabilitation. Each participant must have at least two matched bilateral carious primary molars that require either pulpotomy or indirect pulp cap. Maxillary and mandibular primary first and second molars who receive pulpotomy and /or indirect pulp cap will be compared. The research will be split mouth design where the primary molar on one side will get MTA as the pulpotomy or IPC medicament and the corresponding primary on the other side will get Biodentine as the pulpotomy or IPC medicament in the same arch.

The procedures will be performed according to standards of the American Academy of Pediatric Dentistry (AAPD), by Institutional Review Board approved investigators. Data will be extracted from the electronic health record (EHR) and TigerView dental radiograph imaging software. Data will be recorded using REDCap. Clinical and radiographic follow up of patients will be every 6 months since date of procedure for 3 years. Follow up will be done at the Geisinger Pediatric Dental Clinic at Danville or Milton.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ages of 2 to ≤12 years.
* Bilateral symptomatic or asymptomatic vital primary molars with caries approximating or into the pulp.
* Patient who need a pulpotomy and/or indirect pulp cap treatments in two or more quadrants.
* Parents of patients who can provide consent in English.
* Patients who need treatment in an operating room setting at Geisinger.

Exclusion Criteria:

* Pre-operative radiographic or clinical symptoms associated with irreversible pulpitis or necrotic pulp.
* Radiographs not displaying furcation region of the tooth.
* Patients with cardiac conditions who need prophylaxis for infective Endocarditis.
* Patients with any type of cancer in the past or present.
* Non-restorable molars.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 646 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical success in pulpotomies and indirect pulp caps | 4 years
  To compare the rate of clinical success in primary molars using MTA versus Biodentine in pulpotomies and indirect pulp caps. Subjects will been seen at follow-up standard of care visits every 6 months for 3 years to clinically evaluate if the treatment was successful, if any discoloration has occurred and assess for any signs or symptoms of an abscess.
Rate of radiographic success in pulpotomies and indirect pulp caps | 4 years
  To compare the rate of radiographic success in primary molars using MTA versus Biodentine in pulpotomies and indirect pulp caps. Subjects will been seen at follow-up standard of care visits every 6 months for 3 years where x-rays will be taken to determine if any abscess have formed.

CONTACTS AND LOCATIONS:
Overall Officials: Gayatri Malik, DMD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No